CLINICAL TRIAL: NCT07398651
Title: Comparative Study Between Apremilast and Adalimumab in Psoriatic Arthritis Patients
Brief Title: Apremilast and Adalimumab in Psoriatic Arthritis Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, MenaaAllah Mohamed Elmalla, Assistant Lecturer of Rheumatology, Rehabilitation & Physical Medicine, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 36265MD4108/12 / 25
Record Dates: First submitted 2026-01-29; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Psoriatic Arthritis; Ultrasound Assessment; TNF
Keywords: Psoriatic Arthritis Patients:; Apremilast; Adalimumab
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — Adalimumab; apremilast

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Experimental): consists of 30 PsA patients who will receive Adalimumab with methotrexate therapy for 3 months.
  Interventions: Drug: Adalimumab
- Group II (Experimental): consists of 30 PsA patients who will receive Apremilast with methotrexate therapy for 3 months.
  Interventions: Drug: Apremilast

INTERVENTIONS:
Drug: Adalimumab — PsA patients who will receive Adalimumab with methotrexate therapy for 3 months
  Arms: Group I
Drug: Apremilast — PsA patients who will receive Apremilast with methotrexate therapy for 3 months
  Arms: Group II

SUMMARY:
The aim of this work is to compare the efficacy of Apremilast combined with Methotrexate versus Adalimumab combined with Methotrexate

DETAILED DESCRIPTION:
Psoriatic arthritis is a heterogeneous chronic systemic auto-immune disease, with variable musculoskeletal involvement as well as skin and nail disease . Up to 30% of patients with psoriasis may develop Psoriatic arthritis over the course of their lifetime. Musculoskeletal manifestations of Psoriatic arthritis include peripheral arthritis, spondylitis, dactylitis and enthesitis.

The pathogenesis of Psoriatic arthritis is still unclear, due to the heterogeneity of the pathogenic pathways involved, the variable clinical manifestations, and different responses to treatment.

A predisposing genetic background in the presence of environmental factors, such as infections, microbiota (dysbiosis), obesity, biomechanical stress could activate the immune system and precipitate the onset of the disease.

Objectives:

* Assessment of the effect of the studied drugs on the disease activity clinically and laboratory in PsA patients.
* Assessment of the effect of the studied drugs on functional status of PsA patients.
* Evaluation of the effect of the studied drugs on the musculoskeletal ultrasound findings of PsA patients

Objectives:

* Assessment of the effect of the studied drugs on the disease activity clinically and laboratory in PsA patients.
* Assessment of the effect of the studied drugs on functional status of PsA patients.
* Evaluation of the effect of the studied drugs on the musculoskeletal ultrasound findings of PsA patients

Musculoskeletal ultrasound is considered one of the most important tools in studying the effects of rheumatic diseases on musculoskeletal structures.

It is demonstrated that ultrasound is more sensitive than conventional radiography and clinical examination for the assessment of inflammatory and structural changes in inflammatory arthritis, including Psoriatic arthritis, and particularly synovitis, enthesitis, tenosynovitis, and bursitis.

The treatment of Psoriatic arthritis requires attention to the active domains present in each patient. If the major active domain is peripheral arthritis, treatment usually begins with non-steroidal anti-inflammatory drugs to control symptoms of pain and mild inflammation. If these drugs fail to control disease activity, a conventional synthetic DMARDs is usually prescribed, most commonly methotrexate. Leflunomide and sulfasalazine have also been used in the management of peripheral joint disease. The European Alliance of Associations for Rheumatology guidelines on the management of Psoriatic arthritis with drug therapies suggest that if patients do not attain a satisfactory response

ELIGIBILITY:
Inclusion Criteria:

* This study will include 60 adult Psoriatic arthritis patients >18 years old, fulfilling the (CASPAR) classification criteria of Psoriatic arthritis and have an inadequate response to methotrexate therapy for at least 3 months.

  * Psoriatic arthritis patients with peripheral musculoskeletal domains (peripheral arthritis, dactylitis and enthesitis) as well as skin and nail domains

Exclusion Criteria:

* Patients who received previous biologic agents or Janus kinase inhibitors.
* Patients with axial and ocular involvement.
* Current or recent serious infection including tuberculosis or hepatitis B/C .
* Current or past history of malignancy (within five year).
* Pregnant or breastfeeding women or women planning pregnancy during the study period .
* Severe uncontrolled comorbidities such as heart failure, severe liver disease, or chronic kidney disease (eGFR <30 mL/min/1.73m²) .

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-12-30 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Disease Activity Index for Psoriatic Arthritis | 3 months
  Assessment of disease activity in psoriatic arthritis patients by Disease Activity Index for Psoriatic Arthritis

SECONDARY OUTCOMES:
Health assessment questionnaire disability index | 3 months
  Functional assessment Using health assessment questionnaire disability index
Psoriasis Area and Severity Index | 3 months
  Psoriasis Area and Severity Index (PASI) for skin involvement

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All data ill be available if it needed
Supporting Information: Study Protocol, SAP, ICF